CLINICAL TRIAL: NCT01642615
Title: A Phase 2 Multicenter, 36-Week Study to Assess the Safety and Effectiveness of Daily Oral Administration of Dexlansoprazole Delayed-Release Capsules for Healing of Erosive Esophagitis and Maintenance of Healed Erosive Esophagitis and Relief of Heartburn, in Adolescent Subjects Aged 12 to 17 Years
Brief Title: Safety and Efficacy of Dexlansoprazole Delayed-Release Capsules for Healing of Erosive Esophagitis and Maintenance of Healed Erosive Esophagitis and Relief of Heartburn in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-390MR_207; U1111-1128-6117 (Registry Identifier: WHO); 2012-001681-15 (EudraCT Number)
Record Dates: First submitted 2012-07-12; First posted 2012-07-17 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Gastroesophageal Reflux Disease; Erosive Esophagitis
Keywords: Drug therapy
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Dexlansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healing Phase: Dexlansoprazole 60 mg (Experimental): Dexlansoprazole 60 mg delayed-release capsules, orally, once daily for up to 8 weeks.
  Interventions: Drug: Dexlansoprazole
- Maintenance Phase: Dexlansoprazole 30 mg (Experimental): Participants who are healed at Week 8 will be randomized to receive 30 mg dexlansoprazole delayed-release capsules, orally, once daily for up to 16 weeks.
  Interventions: Drug: Dexlansoprazole
- Maintenance Phase: Placebo (Experimental): Participants who are healed at Week 8 will be randomized to receive dexlansoprazole placebo-matching capsules, orally, once daily for up to 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexlansoprazole — Dexlansoprazole capsules
  Other Names: Dexilant
  Arms: Healing Phase: Dexlansoprazole 60 mg
Drug: Dexlansoprazole — Dexlansoprazole capsules
  Other Names: Dexilant
  Arms: Maintenance Phase: Dexlansoprazole 30 mg
Drug: Placebo — Dexlansoprazole placebo-matching capsules
  Arms: Maintenance Phase: Placebo

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of treatment with once daily oral administration of dexlansoprazole delayed-release capsules in adolescents with erosive esophagitis (EE) and for maintenance of healed EE and relief of heartburn.

DETAILED DESCRIPTION:
The drug being tested in this study is called dexlansoprazole. Dexlansoprazole is being tested to treat adolescents who have erosive esophagitis and heartburn and maintenance of healing of EE.

The study planned to enroll approximately 60 patients.

The study consisted of 3 periods:

1. Screening ((21 [+5] days)
2. Treatment (8 weeks for healing, 16 weeks for maintenance),
3. Post-Treatment Follow-up (up to 3 months).

During screening, participants used an electronic diary (eDiary) daily to document the presence of daytime and nighttime heartburn symptoms and the degree to which heartburn hurt (hereinafter referred to as severity), and to record their use of rescue medication (antacid).

During the first 8 week treatment period, all participants received dexlansoprazole 60 mg, once daily (QD). At the Week 8 visit, participants underwent endoscopy to assess healing of EE. Participants whose EE had not healed were discontinued from the study.

Participants whose EE had healed were randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* dexlansoprazole 30 mg QD
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient

All participants were asked to take one tablet each morning without regard to food throughout the study. Throughout both phases of the Treatment Period, all participants continued to use the eDiary to document the presence or absence and severity of daytime and nighttime heartburn symptoms and the use of rescue medication.

This multi-center trial was conducted worldwide. The overall time to participate in this study was 39 weeks. Participants made multiple visits to the clinic, and were contacted by telephone during the study

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant and parent(s) or legal guardian are capable of understanding and complying with protocol requirements.
2. Prior to any study-specific procedures being performed, the informed consent and the assent form, according to local country requirements, must be signed and dated by parent(s) or legal guardian and by the participant respectively.
3. The participant has a medical history of symptoms of Gastroesophageal Reflux Disease (GERD) for at least 3 months prior to Screening (signed informed consent form and assent, if applicable) as assessed by the investigator.
4. The participant has met the electronic diary qualification criteria as assessed by the electronic daily diary defined as follows: heartburn (burning or hurting in your throat, chest, or stomach) on at least 3 of 7 days.(Note: if an endoscopy done within 1 week of signing informed consent and assent is used to confirm diagnosis of EE, the subject does not need to meet this criterion).
5. The participant has endoscopic evidence of EE (LA Grade A-D) based on the screening endoscopy.
6. The participant is male or female and aged 12 to 17 years, inclusive.
7. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent and assent throughout the duration of the study and for 30 days after last dose of study medication.
8. A female participant of childbearing potential who is or may become sexually active agrees to routinely use adequate contraception from the time of signing the informed consent and assent until 30 days after the last dose of study medication.

Exclusion Criteria:

1. Participant has evidence of cardiovascular, pulmonary, central nervous system, hepatic, hematopoietic, renal, metabolic, endocrine or gastrointestinal disease, or serious allergy, asthma, or allergic skin rash that suggests clinically significant, uncontrolled underlying disease or condition (other than the disease being studied), which may impact the ability of the participant to participate or potentially confound the study results.
2. The participant has a co-existing disease affecting the esophagus (eg, esophageal varices, scleroderma, viral or fungal infection, or esophageal stricture), history of radiation therapy or cryotherapy to the esophagus, caustic or physiochemical trauma such as sclerotherapy to the esophagus.
3. The participant has known history of Barrett's with dysplastic changes in the esophagus.
4. The participant has a known history of eosinophilic esophagitis (EoE) or endoscopic findings suggestive of EoE.
5. The participant has a history of celiac disease or participant tests positive for tissue transglutaminase (tTG) antibody.
6. The participant has active gastric or duodenal ulcers within 4 weeks prior to Day -1.
7. Participant has any finding in his/her medical history, physical examination, or safety clinical laboratory tests giving reasonable suspicion of underlying disease that might interfere with the conduct of the trial.
8. Participant has taken any proton pump inhibitor (PPI) within 1 week (7 days) prior to the Screening Visit.
9. Participant tests positive for H. pylori.
10. The participant has a history of hypersensitivity or allergies to dexlansoprazole or any component of dexlansoprazole or any PPI (including lansoprazole, omeprazole, rabeprazole, pantoprazole, or esomeprazole) or antacid containing Mg(OH)2 and/or Al(OH)3 or simethicone.
11. The participant is required to take excluded medications or it is anticipated that the participant will require treatment with at least one of the disallowed concomitant medications during the study evaluation period as specified in the Excluded Medications and Treatments Section 7.3.
12. The participant has a history of malignant disease (except basal cell carcinoma) within 5 years prior to Screening.
13. The participant has a condition that may require inpatient surgery during the course of the study.
14. The participant requires dilatation of esophageal strictures and/or strictures preventing passage of the endoscope during the Screening endoscopy. Schatzki's ring (a ring of mucosal tissue near the lower esophageal sphincter) is acceptable.
15. The participant is known to be human immunodeficiency virus (HIV) positive.
16. The participant has current or clinical history of Zollinger-Ellison syndrome or other hypersecretory condition.
17. The participant has a history of gastric, duodenal or esophageal surgery except simple oversew of an ulcer. A history of gastric tube and/or percutaneous endoscopic gastrostomy (PEG) placement is allowed.
18. The participant had an acute upper gastrointestinal hemorrhage within 4 weeks prior to endoscopy.
19. The participant has donated or lost ≥300 mL blood volume, undergone plasmapheresis, or has had a transfusion of any blood product within 90 days prior to the first dose of study drug.
20. The participant has a known history of alcohol abuse or illegal drug use within the past 12 months prior to the first dose of study drug.
21. The participant has any Screening Visit 1 abnormal laboratory value that suggests a clinically significant underlying disease or condition that may prevent the participant from entering the study; or the participant has: creatinine >1.5 mg/dL, alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2 times the upper limit of normal (×ULN), or total bilirubin >2.0 mg/dL with AST/ALT elevated above the limits of normal values.
22. If female, the participant is pregnant or lactating or intending to become pregnant before, during or within 30 days after last dose of study medication; or intending to donate ova during such time period.
23. If male, the participant intends to donate sperm during the course of this study or within 30 days after last dose of study drug.
24. The participant, participant's Parent(s) or Legal Guardian is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study or may consent and assent under duress. Students of the institution/research facility who are under the supervision of, or in a subordinate role to, the investigator are also ineligible.
25. The participant or participant's Parent(s) or Legal Guardian, in the opinion of the investigator, is unlikely to comply with the protocol requirements or is unsuitable for any other reason.
26. The participant has participated in another clinical study and/or has received any investigational compound within 30 days prior to Screening.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2012-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda Global Research and Development Center, Inc.
Locations (60):
- United States (32):
  - Huntsville, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Los Angeles, California
  - San Francsco, California
  - Centennial, Colorado
  - Thornton, Colorado
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Flint, Michigan
  - Plymouth, Minnesota
  - Jackson, Mississippi
  - Kansas City, Missouri
  - Mays Landing, New Jersey
  - Brooklyn, New York
  - Toledo, Ohio
  - Youngstown, Ohio
  - Greenville, South Carolina
  - Kingsport, Tennessee
  - Fort Worth, Texas
  - Houston, Texas
  - Laredo, Texas
  - San Antonio, Texas
  - Ogden, Utah
  - Salt Lake City, Utah
  - Fairfax, Virginia
  - Norfolk, Virginia
- Brussels, Belgium
- Brazil (4):
  - Passo Fundo, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Santo André, São Paulo
  - São José do Rio Preto, São Paulo
- Hungary (5):
  - Debrecen
  - Győr
  - Miskolc
  - Nyíregyháza
  - Pécs
- Italy (3):
  - Bari, Bari
  - Messina, Messina
  - Roma, Roma
- Mexico (3):
  - Mexico City, Mexico City
  - Monterrey, Nuevo León
  - Culiacán, Sinaloa
- Poland (7):
  - Bydgoszcz
  - Krakow
  - Rzeszów
  - Szczecin
  - Torun
  - Warsaw
  - Wroclaw
- Portugal (5):
  - Amadora
  - Braga
  - Coimbra
  - Lisbon
  - Porto

REFERENCES:
- See also: Dexilant Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=9efb34b3-fb69-4190-a2be-a90b8cb94e25&filetypecode=DEXILANTPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 18 investigative sites in Mexico, Poland, Portugal and the United States from 22 June 2012 (first participant to sign the informed consent) to 10 November 2014.
Pre-assignment Details: Sixty three adolescents with a diagnosis of erosive esophagitis (EE) were enrolled in the dexlansoprazole delayed release 60 mg capsules open label phase. One participant was not treated. Participants with healed EE were randomized into one of 2 treatment groups: dexlansoprazole delayed release 30 mg capsules or placebo in the maintenance phase.
Period: Open Label Maintenance Phase
Arm/Group | Healing Phase: Dexlansoprazole 60 mg | Maintenance Phase: Dexlansoprazole 30 mg | Maintenance Phase: Placebo
Started | 63 | 0 | 0
Safety Analysis Set | 62 | 0 | 0
Completed | 58 | 0 | 0
Not Completed | 5 | 0 | 0
Not completed — Pretreatment Event/Adverse Event | 1 | 0 | 0
Not completed — Major Protocol Deviation | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Voluntary Withdrawal | 1 | 0 | 0
Not completed — Did not receive treatment | 1 | 0 | 0
Period: Double Blind Maintenance Phase
Arm/Group | Healing Phase: Dexlansoprazole 60 mg | Maintenance Phase: Dexlansoprazole 30 mg | Maintenance Phase: Placebo
Started | 0 | 25 | 26
Completed | 0 | 18 | 20
Not Completed | 0 | 7 | 6
Not completed — Lack of Efficacy | 0 | 1 | 3
Not completed — Voluntary Withdrawal | 0 | 5 | 2
Not completed — Pretreatment Event/Adverse Event | 0 | 1 | 0
Not completed — Requires Treatment with Another Drug | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline measures are based on the Safety Analysis Set and included all enrolled participants who received at least one dose of study drug.
Groups:
- All Participants: Dexlansoprazole 60 mg delayed-release capsules, orally, once daily for up to 8 weeks in the Open Label Healing Phase. Participants with healing of EE were eligible to participate in the Maintenance Phase.
Arm/Group | All Participants
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.8 (1.64)
Age, Customized [Number; unit: participants]
  12 to 14 years | 24
  15 to 17 years | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 38
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 16
  Hispanic or Latino | 6
  Not Collected outside the United States | 40
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1
  White | 61
Region of Enrollment [Number; unit: participants]
  United States | 22
  Portugal | 4
  Poland | 34
  Mexico | 2
Height [Mean (Standard Deviation); unit: cm] | 165.5 (9.68)
Weight [Mean (Standard Deviation); unit: kg] | 61.86 (17.060)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI is calculated using the weight and height.
  kg/m^2 | 22.34 (5.086)
Smoking Classification [Number; unit: participants]
  Never smoked | 61
  Current smoker | 1
  Ex-smoker | 0
Helicobacter pylori (H. pylori) Status [Number; unit: participants]
  Positive | 0
  Negative | 61
  Unknown | 1
Erosive Esophagitis Present [Number; unit: participants]
  Yes | 62
  No | 0
Baseline EE Grade (LA Classification) [Number; unit: participants] — A=1 (or more) mucosal break 5 mm or less that does not extend between the tops of two mucosal folds, B=1 (or more) mucosal break more than 5 mm-long that does not extend between the tops of two mucosal folds, C=1 (or more) mucosal break that is continuous between the tops of two or more mucosal folds but that involves less than 75% of the circumference and D=1 (or more) mucosal break that involves at least 75% of the esophageal circumference.
  participants
    A | 34
    B | 26
    C | 1
    D | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience Each Treatment Emergent Adverse Event Experienced by ≥5% of Participants During the 8-week Healing Treatment Period
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A Treatment Emergent Adverse Event (TEAE) is defined as an Adverse Event (AE) that starts or worsens on or after Study Day 1, and no more than 30 days after the last dose.
Time Frame: 8 weeks
Population: Safety analysis set includes all enrolled participants who received at least one dose of open-label study drug in the first 8 weeks.
Measure: Number; unit: percentage of participants
Arm/Group | Healing Phase: Dexlansoprazole 60 mg
Number analyzed (Participants) | 62
percentage of participants
  Diarrhoea | 6.5
  Nasopharyngitis | 6.5
  Headache | 12.9
  Oropharyngeal pain | 8.1

2. Primary Outcome: Percent of Participants Who Experience Each Treatment Emergent Adverse Event Experienced by ≥5% of Participants During the 16-week Maintenance Treatment Period
Description: as for outcome 1
Time Frame: From Week 8 to Week 24
Population: Safety Analysis Set included all participants with healed EE at Week 8 who were randomized and received at least one dose of open-label study drug in Weeks 8 to 24.
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance Phase: Dexlansoprazole 30 mg | Maintenance Phase: Placebo
Number analyzed (Participants) | 25 | 26
percentage of participants
  Abdominal pain | 12.0 | 11.5
  Abdominal pain upper | 4.0 | 7.7
  Erosive oesophagitis | 4.0 | 7.7
  Diarrhoea | 0.0 | 7.7
  Pyrexia | 0.0 | 7.7
  Nasopharyngitis | 12.0 | 15.4
  Pharyngitis | 12.0 | 0.0
  Sinusitis | 12.0 | 0.0
  Upper respiratory tract infection | 8.0 | 0.0
  Bronchitis | 8.0 | 3.8
  Headache | 24.0 | 15.4
  Insomnia | 8.0 | 0.0

3. Secondary Outcome: Percentage of Participants With Healing of Erosive Esophagitis (EE) by Week 8
Description: Healing of EE was assessed by endoscopy.
Time Frame: 8 weeks
Population: Participants from the Full Analysis Set, all enrolled participants who received at least one dose of open-label study drug in the first 8 weeks, with data available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Healing Phase: Dexlansoprazole 60 mg
Number analyzed (Participants) | 58
percentage of participants | 87.9 [76.7 to 95.0]

4. Secondary Outcome: Percentage of Participants Who Maintain Healing of EE From Week 8 to Week 24
Description: Percentage of participants who maintain healing of EE from Week 8 to Week 24 among the patients who were healed at Week 8 as assessed by endoscopy.
Time Frame: From Week 8 to Week 24
Population: Participants from the Full Analysis Set, all participants with healed EE at Week 8 who were randomized and received at least one dose of open-label study drug in Weeks 8 to 24.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Dexlansoprazole 30 mg | Maintenance Phase: Placebo
Number analyzed (Participants) | 22 | 24
percentage of participants | 81.8 [59.7 to 94.8] | 58.3 [36.6 to 77.9]

5. Secondary Outcome: Percent of Days With Neither Daytime Nor Nighttime Heartburn Over the First 8 Weeks of Treatment
Description: Percent of days with neither daytime nor nighttime heartburn over the first 8 weeks of treatment as assessed by electronic daily diary. The percent of days with neither daytime or nighttime heartburn = (total number of days that are heartburn free)/(total number of days for which either a daytime or nighttime result is marked) x 100%.
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent of days
Arm/Group | Healing Phase: Dexlansoprazole 60 mg
Number analyzed (Participants) | 62
percent of days | 59.6 (30.46)

6. Secondary Outcome: Percent of Days With Neither Daytime Nor Nighttime Heartburn Over Weeks 8 to 24
Description: The percent of days with neither daytime nor nighttime heartburn over Weeks 8 to 24 as assessed by electronic daily diary among the participants who were healed at Week 8. The percent of days with neither daytime or nighttime heartburn = (total number of days that are heartburn free)/(total number of days for which either a daytime or nighttime result is marked) x 100%.
Time Frame: Weeks 8 to 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent of days
Arm/Group | Maintenance Phase: Dexlansoprazole 30 mg | Maintenance Phase: Placebo
Number analyzed (Participants) | 24 | 26
percent of days | 76.7 (29.82) | 68.9 (26.04)

ADVERSE EVENTS:
Time Frame: Up to 24 Weeks
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Healing Phase: Dexlansoprazole 60 mg | Maintenance Phase: Dexlansoprazole 30 mg | Maintenance Phase: Placebo
Serious Adverse Events (participants affected / at risk) | 1/62 | 2/25 | 1/26
Other Adverse Events (participants affected / at risk) | 24/62 | 14/25 | 11/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healing Phase: Dexlansoprazole 60 mg (N=62) | Maintenance Phase: Dexlansoprazole 30 mg (N=25) | Maintenance Phase: Placebo (N=26)
Substance abuse (Psychiatric disorders) | 1 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Healing Phase: Dexlansoprazole 60 mg (N=62) | Maintenance Phase: Dexlansoprazole 30 mg (N=25) | Maintenance Phase: Placebo (N=26)
Headache (Nervous system disorders) | 8 | 6 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 2
Nasopharyngitis (Infections and infestations) | 4 | 3 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2
Bronchitis (Infections and infestations) | 1 | 2 | 1
Pharyngitis (Infections and infestations) | 3 | 3 | 0
Sinusitis (Infections and infestations) | 1 | 3 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.